CLINICAL TRIAL: NCT02926820
Title: Working Memory Training in Individuals With Huntington's Disease: A Pilot Project
Brief Title: Working Memory Training in Huntington's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: York University (Other)
Collaborators: North York General Hospital (Other)
Responsible Party: Principal Investigator, Christine Till, Associate Professor, Department of Psychology, York University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NYGH 15-0001
Record Dates: First submitted 2016-09-30; First posted 2016-10-06 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-10

CONDITIONS: Huntington's Disease
Keywords: Huntington disease; cognitive rehabilitation; cognitive dysfunction
MeSH Terms: conditions — Huntington Disease; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cognitive training (Experimental): Participants will undergo five weeks of cognitive training using the Cogmed QM program. All patients complete the same intervention.
  Interventions: Behavioral: Cogmed QM

INTERVENTIONS:
Behavioral: Cogmed QM — The intervention consisted of 25 Cogmed sessions, typically completed over a five week period (i.e. 5 days per week), with each session lasting between 40-50 minutes per day. The program consists of 12 exercises that target visuo-spatial or verbal working memory. At each training session, participants completed 8 of the 12 exercises (order selected by the user), with 15 trials per exercise. Cogmed QM is an adaptive program, wherein task difficulty is adjusted to performance on each trial. The level of difficulty adjusts continuously and automatically, ensuring that each session provides an engaging, challenging level of WM capacity. Breaks were permitted, and encouraged, at the participants' discretion throughout the session.

SUMMARY:
There is a paucity of investigation into effective interventions to enhance cognitive function and/or mitigate cognitive decline in individuals with Huntington disease (HD). This study targeted working memory (WM), which is the ability to actively hold information in the mind in order to perform complex mental tasks, given reports of WM dysfunction in patients with HD. The investigators examined the feasibility of conducting a 5-week WM training program (Cogmed). Patient adherence and treatment tolerance were assessed. In addition, preliminary evidence for the efficacy of this training program on targeted cognitive abilities was examined. Nine patients with pre-manifest or early stage HD underwent training. Patients were assessed before the intervention and one week after completion.

DETAILED DESCRIPTION:
Huntington disease (HD) is associated with a variety of cognitive deficits, with prominent difficulties in working memory (WM). WM deficits are notably compromised in early-onset and prodromal HD patients. This study aimed to determine the feasibility of a computer-ized WM training program (Cogmed QM), novel to the HD population. Nine patients, aged 26-62, with early stage HD underwent a 25-session (5 days/week for 5 weeks) WM training program (Cogmed QM). Training exercises involved the manipulation and storage of verbal and visuospatial information, with difficulty adapted as a function of individual performance. Neuropsychological testing was conducted before and after training, and performance on criterion WM measures (Digit Span and Spatial Span) and near-transfer WM measures (Symbol Span and Auditory WM) were evaluated. Post-training inter-views about patient experience were thematically analyzed using NVivo software. Seven of nine patients demonstrated adherence to the training and completed all sessions within the recommended timeframe of 5 weeks. All adherent patients reported that they found training helpful (n=7), and almost all felt that their memory improved (n=6). Compared to baseline scores, patients showed significant improvement on the neuropsychological measures of verbal WM, including Digit Span (p = .047) and Auditory WM (p = .041). This pilot study provides support for feasibility of computerized WM training in early-stage patients with HD. Results suggest that HD patients can improve WM with intensive training, though a full-scale intervention project is needed to understand the reliability of changes over time.

ELIGIBILITY:
Inclusion Criteria:

1. Laboratory-confirmed gene expansion of at least 36 CAG repeats
2. Reported working memory difficulties on the Patient-Reported Outcomes in Cognitive Impairment (PROCOG) questionnaire
3. Total Functional Capacity (TFC) score of at least 3, taken from the UHDRS
4. Montreal Cognitive Assessment (MOCA) score of 19 or greater

Exclusion Criteria:

1. History of head trauma/neurological event such as stroke
2. Untreated psychiatric symptoms or substance abuse
3. Visual or motor symptoms that would impede ability to complete the program and/or neuropsychological testing
4. Nonfluency in English

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-02; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Adherence to training (defined by completing the intervention within the recommended time frame) | 40 days
  Adherence was defined as completion of at least 80% of the total 25 training sessions within 40 calendar days or less

SECONDARY OUTCOMES:
Digit Span subtest from the Wechsler Memory Scales - third edition | Baseline (time 0) versus Post-intervention test score (up to 45 days post-baseline)
  This test is used as a criterion measure (i.e. measure that closely resembles tasks in the Cogmed program). Scores will be reported in raw score units as the total correct responses.
Spatial Span subtest from the Wechsler Memory Scales - third edition | Baseline (time 0) versus Post-intervention test score (up to 45 days post-baseline)
  This test is used as a criterion measure (i.e. measure that closely resembles tasks in the Cogmed program). Scores will be reported in raw score units as the total correct responses.
Auditory Working Memory from the Woodcock Johnson Tests of Cognitive Ability - third edition | Baseline (time 0) versus Post-intervention test score (up to 45 days post-baseline)
  This test is used as a near transfer measure (i.e. test of verbal or visuospatial working memory that include stimuli that are similar to trained tasks). Scores will be reported in raw score units (total correct responses)
Symbol span subtest from the Wechsler Memory Scales - fourth edition, reported in raw score units (total correct responses) | Baseline (time 0) versus Post-intervention test score (up to 45 days post-baseline)
  This test is used as a near transfer measure (i.e. test of verbal or visuospatial working memory that include stimuli that are similar to trained tasks). Scores will be reported in raw score units (total correct responses)
Verbal Fluency subtest from the Delis-Kaplan Executive Function System | Baseline (time 0) versus Post-intervention test score (up to 45 days post-baseline)
  This tests is used as a control task (i.e tests that do not directly assess working memory). Score will be reported in raw score units (total words produced)
Symbol Digits Modalities Test (oral administration) | Baseline (time 0) versus Post-intervention test score (up to 45 days post-baseline)
  This tests is used as a control task (i.e tests that do not directly assess working memory). Score will be reported in raw score units (total words produced)
Word List Learning from the Hopkins Verbal Learning Test -Revised | Baseline (time 0) versus Post-intervention test score (up to 45 days post-baseline)
  This tests is used as a control task (i.e tests that do not directly assess working memory). Score will be reported in raw score units (total words learned)
Trail Making Test - Parts A and B | Baseline (time 0) versus Post-intervention test score (up to 45 days post-baseline)
  This tests is used as a control task (i.e tests that do not directly assess working memory). Score will be reported in raw score units (total time in seconds)

OTHER OUTCOMES:
Qualitative experiences of training program as reported by the patient | Post-interview follow-up, up to 45 days following baseline visit
  Keywords were used to elicit themes that were indicative of participant attitude and motivation for training
Tolerance (ratio of training time to breaks per day) | Per session and through completion of training program, up to 40 days
  To assess tolerance, the ratio of active training time to breaks per day was examined (Cogmed guidelines suggest at most a 2:1 ratio of active training time and breaks per sessions).
Cogmed Improvement Index | Through completion of training program, up to 40 days
  The Improvement Index represents average improvement over the course of the training. It is calculated automatically by the program by subtracting the Start Index (score on third day of training) from the Max Index (best score throughout training).

CONTACTS AND LOCATIONS:
Overall Officials: Christine Till, PhD, Principal Investigator — York University
Locations (1):
- North York General Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sadeghi M, Barlow-Krelina E, Gibbons C, Shaikh KT, Fung WLA, Meschino WS, Till C. Feasibility of computerized working memory training in individuals with Huntington disease. PLoS One. 2017 Apr 28;12(4):e0176429. doi: 10.1371/journal.pone.0176429. eCollection 2017. PMID 28453532